CLINICAL TRIAL: NCT02248246
Title: Prospective, Multicenter, Observational Study Evaluating Vessel Sealing Utilizing the Harmonic ACE®+7 Shears During Laparoscopic Colectomy
Brief Title: Harmonic ACE®+7 Shears in Laparoscopic Colectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ethicon Endo-Surgery (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ENG-14-001
Record Dates: First submitted 2014-09-22; First posted 2014-09-25 (Estimated); Results first posted 2016-04-01 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-06

CONDITIONS: Benign or Malignant Disease Indicated for Colectomy
Keywords: Hemostasis; Harmonic ACE®+7 Shears; Laparoscopic; Inferior mesenteric artery; Inferior mesenteric vein; Observational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Colectomy with Harmonic ACE®+7 Shears (Other): Laparoscopic colectomy with Harmonic ACE®+7 Shears for dissection and vessel transection
  Interventions: Device: Harmonic ACE®+7 Shears

INTERVENTIONS:
Device: Harmonic ACE®+7 Shears — Vessel sealing performance assessed for transection and sealing of the following named vessels:
  * Inferior mesenteric artery (IMA)
  * Inferior mesenteric vein (IMV) (if identified)

SUMMARY:
This is a prospective, non-randomized, single arm, multicenter, observational study to assess the initial clinical experience with the Harmonic ACE®+7 Shears by evaluating vessel sealing during laparoscopic colectomy. The study will not modify or influence current surgeon technique. Investigators will perform each procedure using the device in compliance with their standard surgical approach and product labeling.

The Harmonic ACE®+7 Shears is cleared for commercial distribution and will be used in accordance with approved product labeling. The Harmonic ACE®+7 Shears will be assembled, calibrated, and/or used in accordance with manufacturer design specifications, product instructions and guidelines.

DETAILED DESCRIPTION:
Study Population: Subjects enrolled into this study will undergo elective laparoscopic colectomy wherein dissection and transection of the (inferior mesenteric artery) IMA is indicated.

Primary Variable: Incidence of hemostasis at the IMA Secondary Endpoint: Incidence of hemostasis at the inferior mesenteric vain (IMV).

Definition: Hemostasis of the IMA and IMV is a dichotomous variable (i.e. yes or no). "Yes" is defined as a single activation of the Advanced Hemostasis Mode to transect and seal the IMA and IMV.

Additional exploratory endpoints include:

The percentage of subjects requiring additional measures to obtain hemostasis on the IMA and/or IMV, if identified:

* Number of Harmonic touch ups - frequency of Harmonic reapplications required due to oozing or bleeding at initial transection of named vessels
* Use of other energy devices (tissue sealers, cautery devices) - Graded as yes or no; if "yes", the type, transection time (using stopwatch), time of application (24 hour clock)
* Use of hemostatic products (e.g. hemoclips, staples, sutures, fibrin sealants) - Graded as yes or no; if "yes", the type and name of product, number/volume, and time of application (24 hour clock)

Summary of the use of additional treatment after first pass hemostasis has already been achieved at the IMA and IMV. Graded as yes or no; if "yes", the type, number/volume, time of application (24 hour clock) and rationale for use.

Adverse events attributed to the study device or procedure will be collected from time of surgery to Visit 4 (Approximately 4 weeks after study surgery or as per standard of care (SOC)).

Sample size: No formal sample size determination is required for this study. Approximately 40 subjects from the United States and the European Union are planned to be enrolled into this study.

Global indication for use of the The Harmonic ACE®+7, 5mm Diameter Shears with Advanced Hemostasis:

Indicated for soft tissue incisions when bleeding control and minimal thermal injury are desired. The instruments can be used as an adjunct to or substitute for electrosurgery, lasers and steel scalpels in general, plastic, pediatric, gynecologic, urologic, thoracic, exposure to orthopedic structures (such as spine and joint space), sealing and transection of lymphatic vessels, and other open and endoscopic procedures. The instruments allow for the coagulation of vessels up to and including 7mm in diameter, using the Advanced Hemostasis function.

ELIGIBILITY:
Inclusion Criteria:

1. Indicated for elective laparoscopic colectomy
2. Planned dissection and transection of the IMA
3. Age: equal to or more than18 years

Exclusion Criteria:

Preoperative exclusion criteria:

1. Known or suspected uncontrolled bleeding disorders
2. Subjects unlikely to comply with protocol procedures or adhere to the study visit schedule
3. Any condition rendering a subject unable to understand the nature, scope, and possible consequences of the study or study procedures, or
4. Any Subject unwilling to sign the study informed consent document

   Intra-operative exclusion criteria:
5. Prior to transection of the IMA, the investigator prospectively concludes the inability to safely isolate and transect the IMA with exclusive use of study device while adhering to the instructions for use, or
6. Any intra-operative findings identified by the surgeon that may preclude conduct of the study procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-08; Primary Completion 2015-02 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (2):
  - Jackson Medical Group, Miami, Florida
  - Colorectal Surgical Associates Ltd, LLP, Houston, Texas
- Ziekenhuis Oost-Limburg, Dept of Surgical Oncology, Genk, Belgium
- The Royal Surrey County Hospital NHS Trust, Guildford, Surrey, United Kingdom

REFERENCES:
- [Background] Plasencia G, Van der Speeten K, Hinoul P, Kelch JA, Batiller J, Severin KS, Schwiers ML, Rockall T. Large-Vessel Sealing in Laparoscopic Colectomy with an Ultrasonic Device. JSLS. 2016 Apr-Jun;20(2):e2016.00010. doi: 10.4293/JSLS.2016.00010. PMID 27186065

RESULTS

PARTICIPANT FLOW:
Groups:
- Colectomy With Harmonic ACE®+7 Shears: Laparoscopic colectomy with Harmonic ACE®+7 Shears for dissection and vessel transection
  Harmonic ACE®+7 Shears: Vessel sealing performance assessed for transection and sealing of the following named vessels:
  * Inferior mesenteric artery (IMA)
  * Inferior mesenteric vein (IMV) (if identified)
Period: Overall Study
Arm/Group | Colectomy With Harmonic ACE®+7 Shears
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Safety Set - all subjects in whom the procedure was started.
Arm/Group | Colectomy With Harmonic ACE®+7 Shears
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.8 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 40
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Belgium | 15
  United States | 14
  United Kingdom | 11

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Hemostasis at the IMA
Description: Hemostasis of the IMA is a dichotomous variable (i.e. yes or no). "Yes" is defined as a single activation of the Advanced Hemostasis Mode to transect and seal the IMA.
Time Frame: Intraoperatively
Population: Safety Set - all subjects in whom the procedure was started.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Colectomy With Harmonic ACE®+7 Shears
Number analyzed (Participants) | 40
percentage of subjects | 100.0 [91.2 to 100.0]

2. Secondary Outcome: Percentage of Participants With Hemostasis at the IMV
Description: Hemostasis of the IMV is a dichotomous variable (i.e. yes or no). "Yes" is defined as a single activation of the Advanced Hemostasis Mode to transect and seal the IMV.
Time Frame: Intraoperatively
Population: Safety Set - all subjects in whom the procedure was started.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Colectomy With Harmonic ACE®+7 Shears
Number analyzed (Participants) | 40
percentage of participants | 97.5 [86.8 to 99.9]

ADVERSE EVENTS:
Arm/Group | Colectomy With Harmonic ACE®+7 Shears
Serious Adverse Events (participants affected / at risk) | 5/40
Other Adverse Events (participants affected / at risk) | 20/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Colectomy With Harmonic ACE®+7 Shears (N=40)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (2)
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 1 (1)
Postoperative ileus (Injury, poisoning and procedural complications) | 2 (2)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Splenic haematoma (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Colectomy With Harmonic ACE®+7 Shears (N=40)
Nausea (Gastrointestinal disorders) | 9
Vomiting (Gastrointestinal disorders) | 4
Pain (General disorders) | 7
Wound infection (Infections and infestations) | 2
Procedural pain (Injury, poisoning and procedural complications) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PIs agreed that the first publication of results should be made in conjunction with the presentation of a joint, multicenter publication of the results with all PIs contributing data, analyses, and comments. If this publication was not submitted within 12 months after conclusion of the Study at all sites, or after Sponsor confirmed there would be no multicenter Study publication, whichever is first, the PIs could have published the results from their individual sites.